CLINICAL TRIAL: NCT01933295
Title: Behavioral Treatment of Menopausal Insomnia; Sleep and Daytime Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christopher Drake (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Wayne State University (Other); University of Michigan (Other)
Responsible Party: Sponsor-Investigator, Christopher Drake, Bioscientific Staff, Henry Ford Health System
Organization: Henry Ford Health System (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NR013959; R01NR013959-01 (NIH)
Record Dates: First submitted 2012-09-06; First posted 2013-09-02 (Estimated); Results first posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Menopause
Keywords: treatment
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sleep Education (Active Comparator): Weekly educational emails sent to participants with information about sleep science and tips for better sleep.
  Interventions: Behavioral: Sleep Education
- Cognitive Behavioral Therapy for Insomnia (Experimental): Behavioral treatment (5 component)
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia
- Sleep Restriction Therapy (Experimental): Brief sleep restriction therapy.
  Interventions: Behavioral: Sleep Restriction Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia
  Arms: Cognitive Behavioral Therapy for Insomnia
Behavioral: Sleep Education
  Arms: Sleep Education
Behavioral: Sleep Restriction Therapy
  Arms: Sleep Restriction Therapy

SUMMARY:
Insomnia is recognized as the most prevalent and "costly" sleep disorders and is associated with considerable morbidity including significantly reduced quality of life, impaired work performance, and increased risk for major depressive disorder.1-4 Insomnia is a key symptom of the menopausal transition. Cognitive-behavioral therapy for insomnia (CBT-I) yields equivalent short-term efficacy and superior long-term durability to pharmacological treatment of insomnia. The efficacy of cognitive behavioral therapy for insomnia comorbid with menopause will be tested.

DETAILED DESCRIPTION:
Specific Aim 1: Determine the efficacy of multi-component CBT-I compared to a wait-list control group on self report and laboratory-based polysomnographic (PSG) sleep parameters. We hypothesize that multicomponent CBT-I will increase sleep efficiency, reduce the frequency of awakenings, reduce wake after sleep onset, and increase sleep bout duration compared to the control group evaluated using polysomnographic (PSG) and self-report measures of sleep.

Specific Aim 2a: Test the efficacy of a brief two week single component sleep restriction therapy (SRT) to a wait-list control group on PSG and self-report sleep measures (sleep efficiency, frequency of awakenings, wake after sleep onset, and sleep bout duration). We hypothesize that brief SRT will be efficacious compared to the control condition in women with menopausal-related insomnia.

Specific Aim 2b: Test the comparability (non-inferiority analysis) of SRT to CBT-I. We hypothesize that SRT will produce comparable efficacy in terms of the PSG and self-report measures of sleep compared to CBT-I (primary endpoints: sleep efficiency, frequency of awakenings, wake after sleep onset, and sleep bout duration).

Specific Aim 3: Determine if CBT-I and SRT improves specific aspects of daytime functioning in patients with menopausal-related insomnia. We hypothesize that patients treated with CBT-I or SRT will have greater improvements in depressive symptomatology, quality of life, sleepiness and fatigue compared with a wait list control group.

ELIGIBILITY:
Inclusion Criteria:

* post-menopausal insomnia

Exclusion Criteria:

* unstable medical conditions

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Drake, PhD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

REFERENCES:
- [Derived] Kalmbach DA, Cheng P, Roth T, Sagong C, Drake CL. Objective sleep disturbance is associated with poor response to cognitive and behavioral treatments for insomnia in postmenopausal women. Sleep Med. 2020 Sep;73:82-92. doi: 10.1016/j.sleep.2020.04.024. Epub 2020 May 7. PMID 32799029
- [Derived] Cheng P, Kalmbach D, Fellman-Couture C, Arnedt JT, Cuamatzi-Castelan A, Drake CL. Risk of excessive sleepiness in sleep restriction therapy and cognitive behavioral therapy for insomnia: a randomized controlled trial. J Clin Sleep Med. 2020 Feb 15;16(2):193-198. doi: 10.5664/jcsm.8164. Epub 2020 Jan 13. PMID 31992407
- [Derived] Kalmbach DA, Cheng P, Arnedt JT, Cuamatzi-Castelan A, Atkinson RL, Fellman-Couture C, Roehrs T, Drake CL. Improving Daytime Functioning, Work Performance, and Quality of Life in Postmenopausal Women With Insomnia: Comparing Cognitive Behavioral Therapy for Insomnia, Sleep Restriction Therapy, and Sleep Hygiene Education. J Clin Sleep Med. 2019 Jul 15;15(7):999-1010. doi: 10.5664/jcsm.7882. PMID 31383238
- [Derived] Kalmbach DA, Cheng P, Arnedt JT, Anderson JR, Roth T, Fellman-Couture C, Williams RA, Drake CL. Treating insomnia improves depression, maladaptive thinking, and hyperarousal in postmenopausal women: comparing cognitive-behavioral therapy for insomnia (CBTI), sleep restriction therapy, and sleep hygiene education. Sleep Med. 2019 Mar;55:124-134. doi: 10.1016/j.sleep.2018.11.019. Epub 2018 Dec 28. PMID 30785053
- [Derived] Drake CL, Kalmbach DA, Arnedt JT, Cheng P, Tonnu CV, Cuamatzi-Castelan A, Fellman-Couture C. Treating chronic insomnia in postmenopausal women: a randomized clinical trial comparing cognitive-behavioral therapy for insomnia, sleep restriction therapy, and sleep hygiene education. Sleep. 2019 Feb 1;42(2):zsy217. doi: 10.1093/sleep/zsy217. PMID 30481333

RESULTS

PARTICIPANT FLOW:
Groups:
- Sleep Education: Weekly educational emails sent to participants with information about sleep science and tips for better sleep.
  Sleep Education
- Cognitive Behavioral Therapy for Insomnia: Behavioral (sleep restriction and stimulus control) and cognitive (eg, cognitive restructuring) components, as well as relaxation strategies (eg, progressive muscle relaxation and autogenic training) and sleep hygiene education.
- Sleep Restriction Therapy: 2-week intervention. Specifically, the initial face-to-face session consisted of reviewing patient sleep history, education and rationale for sleep restriction practices, and behavioral homework. Then four follow-up sessions (three phone contacts, each 3-4 days apart, followed by a second face-to-face session) were delivered across the following 2 weeks and were used to titrate sleep schedules based on sleep diary data.
Period: Overall Study
Arm/Group | Sleep Education | Cognitive Behavioral Therapy for Insomnia | Sleep Restriction Therapy
Started | 50 | 52 | 52
Completed | 43 | 41 | 42
Not Completed | 7 | 11 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sleep Education | Cognitive Behavioral Therapy for Insomnia | Sleep Restriction Therapy | Total
Number analyzed (Participants) | 50 | 52 | 52 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.24 (5.55) | 55.32 (5.90) | 56.76 (5.39) | 56.44 (5.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 52 | 52 | 154
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 20 | 22 | 17 | 59
  White | 26 | 24 | 28 | 78
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 3 | 6 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Diary Based Sleepiness
Description: Diaries were based on the consensus sleep diaries but were modified to also measure patient sleepiness over the past 24 hours on a 0 "none" to 10 "highest" scale. Scores in this study represent the daily mean for sleepiness ratings for each assessment period: "pre-treatment (baseline), post-treatment (approximately 4 weeks after baseline), and 6 month follow-up (approximately 7-8 months after baseline)
Time Frame: 8 months
Population: Lost to follow-up at 6 months follow-up assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sleep Education | Cognitive Behavioral Therapy for Insomnia | Sleep Restriction Therapy
Number analyzed (Participants) | 50 | 52 | 52
score on a scale
  Pre Treatment | 5.01 (1.65) | 5.13 (1.68) | 4.87 (1.70)
  Post Treatment | 4.72 (2.06) | 4.36 (2.16) | 4.09 (2.07)
  6 months follow up: number analyzed (Participants) | 43 | 41 | 42
  6 months follow up | 4.73 (1.97) | 3.43 (1.90) | 3.47 (2.04)

2. Secondary Outcome: Fatigue Severity Scale (FSS).
Description: Scores range from 9 to 63, with higher scores indicating greater fatigue, and scores above 36 indicate severe fatigue.
  Data collected at pre-treatment (baseline), post-treatment (approximately 4 weeks after baseline), and 6 month follow-up (approximately 7-8 months after baseline).
Time Frame: 8 months
Population: Lost to follow-up at 6 months follow-up assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sleep Education | Cognitive Behavioral Therapy for Insomnia | Sleep Restriction Therapy
Number analyzed (Participants) | 50 | 52 | 52
score on a scale
  Pre Treatment | 32.50 (11.68) | 31.78 (10.89) | 33.28 (11.68)
  Post Treatment | 32.32 (11.95) | 28.20 (10.32) | 29.90 (12.08)
  6 months follow-up: number analyzed (Participants) | 43 | 41 | 42
  6 months follow-up | 32.31 (10.95) | 25.35 (10.41) | 28.49 (10.74)

3. Secondary Outcome: Medical Outcomes Study Short Form Health Survey (SF-36), Energy Subscale
Description: Domain scores range from 0 to 100 with higher scores indicating better quality of life.
  Data collected at each assessment period: "pre-treatment (baseline), post-treatment (approximately 4 weeks after baseline), and 6 month follow-up (approximately 7-8 months after baseline)
Time Frame: 8 months
Population: Lost to follow-up at 6 months follow-up assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Cognitive Behavioral Therapy for Insomnia: Behavioral treatment (5 component)
  Cognitive Behavioral Therapy for Insomnia
- Sleep Restriction Therapy: Brief sleep restriction therapy.
  Sleep Restriction Therapy
Arm/Group | Sleep Education | Cognitive Behavioral Therapy for Insomnia | Sleep Restriction Therapy
Number analyzed (Participants) | 50 | 52 | 52
score on a scale
  Pre-Treatment | 52.70 (19.51) | 52.50 (18.11) | 52.76 (21.02)
  Post-Treatment | 52.10 (19.77) | 61.90 (18.07) | 61.33 (17.76)
  6 months follow-up: number analyzed (Participants) | 43 | 41 | 42
  6 months follow-up | 54.55 (19.10) | 67.79 (16.49) | 65.70 (17.48)

ADVERSE EVENTS:
Time Frame: Through study completion, consisting of 8 months of study participation for each participant.
Description: The definition of adverse event and/or serious adverse event, used to collect adverse event information, doesn't differ from the clinicaltrials.gov definitions.
Arm/Group | Sleep Education | Cognitive Behavioral Therapy for Insomnia | Sleep Restriction Therapy
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 0/50 | 0/52 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-04-19): https://cdn.clinicaltrials.gov/large-docs/95/NCT01933295/Prot_SAP_000.pdf
  • Informed Consent Form (2017-04-19): https://cdn.clinicaltrials.gov/large-docs/95/NCT01933295/ICF_001.pdf